CLINICAL TRIAL: NCT05591963
Title: Determination of Pre- and Post-Operational Nutritional Status in Orthognathic Surgery Patients
Brief Title: Nutritional Status in Orthognathic Surgery Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MU_DHF_SBF_02
Record Dates: First submitted 2022-09-29; First posted 2022-10-24 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Malocclusion
Keywords: Orthognathic surgery; Malocclusion; Nutritional Status
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the effect of orthognathic surgery on nutritional status, anthropometric measurements, food consumption levels, physical activity levels, biochemical parameters, chewing ability and oral-health impact profile.

DETAILED DESCRIPTION:
Sub-objectives of the study;

* Determining nutritional status changes after orthognathic surgery
* Determining changes in anthropometric measurements (body weight, BMI, fat mass, muscle mass, total body water, waist circumference, hip circumference, mid-upper arm circumference) after orthognathic surgery
* Determining food consumption changes after orthognathic surgery
* Determining changes is physical activity levels after orthognathic surgery
* Determining changes in biochemical parameters 3 months after orthognathic surgery
* Determining changes in chewing ability after orthognathic surgery
* Determining changes in oral-health impact profile after orthognathic surgery
* Determining changes in pain intensity

The aim of this study is to compare these parameters preoperative to postoperative timeline of orthognathic surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old,
* Volunteer to participate in the study,
* Dysgnatic patients with malocclusion who applied to Marmara University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery will be included in the study.
* Type of surgery (only patients with genioplasty operation will not be accepted)

Exclusion Criteria:

* Patients with a history of acute facial trauma,
* Patients with previous facial surgeries,
* Pregnant or lactating women
* Those who have diseases that may cause systemic neuropathy such as diabetes, hypertension, kidney disease,
* Those who do not want to sign the consent form,
* Orthognathic surgery patients treated with genioplasty only,
* Patients with a history of eating disorders (anorexia nervosa, bulimia nervosa, etc.).
* Patients with a history of malignancy, radiotherapy or chemotherapy will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who applied to the Marmara University Faculty of Dentistry Department of Oral and Maxillofacial Surgery who applied for dentomaxillofacial deformities and needed orthognathic surgery will be included in the study. It is aimed to invite all patients who applied to the clinic to the research.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in nutritional status | 3 months
  The Subjective Global Assessment (SGA) will be used to assess changes in nutritional status. SGA is an easy-to-apply, low-cost and reliable method that is frequently used in the evaluation of malnutrition status. After the patient is evaluated according to certain criteria, the level of malnutrition is determined by the evaluator's subjective point of view. It is a four-part evaluation. These are weight loss and food intake history, gastrointestinal system symptoms, functional capacity, metabolic requirement, and physical examination. The analysis of the information and the results from it are scored as A, B, C. If the patient is well-nourished, he is classified as A, moderately malnourished, B, and severely malnourished, C. SGA will be applied by the researchers in face-to-face meetings within 7 days before the operation, on the 7th day, 15th day, 1st month and 3rd month after the operation.
Change in food consumption | 3 months
  To evaluate the food consumption of the patients included in the study, at the preop 7 days, postoperative 7th day, 15th day, 1st month and 3rd month will be taken with 24-hour recall method. The amount of nutrients included in the meals will be calculated by using the "Standard Recipes" book, and the measurement amounts will be calculated by using the "Food Photo Catalogue" book. The data obtained from the 24-hour recall method will be analyzed using the "Computer Assisted Nutrition Program, Nutrition Information Systems Package Program (BEBIS)" and the amount of energy, carbohydrates, protein, fat, fiber and micronutrients consumed by participants will be calculated. Intake of energy, macro nutrients, fiber and micronutrients will be compared with the preop 7 days, postoperative 7th day, 15th day, 1st month and 3rd.
Change in chewing ability | 3 months
  In this study, a questionnaire consisting of open and closed-ended questions will be used to determine the chewing difficulties of individuals. With open-ended questions, foods that are difficult to chew and the methods used to consume these foods will be questioned. In the follow-up interviews, closed-ended questions such as the ability to chew the previously listed foods are "easy to chew", "I have a little difficulty", "I have a lot of difficulty / can't chew at all". If individuals say, "I have a little or a lot of difficulty" while chewing hard foods and "I have some or a lot of difficulty" when chewing soft foods, they will be evaluated as "difficulty in chewing".
Change in body weight | 3 months
  Body weight will be evaluated during face-to-face interviews with patients in pre-op 7 days and post-op 7th day, 15th day, 1st month and 3rd month with Tanita DC-360 body analyzer. Patients will be asked to remove all metal items (rings, earrings, bracelets, watches, phones, etc.), any heavy clothing, shoes, or socks before stepping on the device. The device was set to -1.0 kg for the remaining clothes.
Change in BMI | 3 months
  Body Mass Index will be calculated as weight (kg)/height (m2) and will be classified based on the WHO classification. It will be evaluated at pre-op 7 days and post-op 7th day, 15th day, 1st month and 3rd month.
Change in Body Composition | 3 months
  Body composition analysis will be performed with the Tanita DC-360 device that performs bioelectrical impedance analysis (BIA). The analysis report includes body weight (kg), body water mass (kg), body fat mass (kg) and body muscle mass (kg). This method is non-invasive and provides body composition data in less than 1 minute of measurement. Using this device, the body compositions of the individuals will be recorded in the pre-op 7 days and on the post-op 7th day, 15th day, 1st month and 3rd month.

SECONDARY OUTCOMES:
Change in physical activity | 3 months
  The pre-op and post-op physical activity levels of the patients included in the study will be evaluated with the short version of the International Physical Activity Questionnaire (IPAQ), which will be administered at each interview. The International Physical Activity Questionnaire Short Version (7 questions) is used for seven days to assess physical activity in 4 domains, including leisure, indoor, work and transport-related physical activity. Physical activity level is classified as active, mildly active and active according to general scores.
Change in Oral-Health Impact Profile | 3 months
  A scale of 1 to 5 will be used to rate each of the 14 questions about how dental health affects quality of life (minimum score of 0, maximum score of 70). Higher ratings reflect a greater influence of the patient's dental health on their quality of life (higher scores, worse outcomes). At baseline and 3rd month of post-op, the questionnaire will be taken.
Change in pain intensity | 3 months
  Change in muscle pain intensity was assessed using a Visual Analogue Scale (VAS) ranging from the absence of pain (score 0) to the most severe pain imaginable. The VAS consist of a line which can be presented horizontally or vertically (10 cm long) with anchor points of "no pain" and "worst possible pain". The patient will be asked to put a mark on the line that best describe the pain severity. The patients' responses' will be recorded and scored according to the VAS scale. Then, the results will be compared with the baseline, 1 month and 6 months later.
Change in Body Circumference Measurements | 3 months
  Waist circumference, hip circumference, upper middle arm circumference will be evaluated during face-to-face interviews with patients in pre-op 7 days and post-op 7th day, 15th day, 1st month and 3rd month. It will be done by the researcher, using international standards for anthropometric measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)